CLINICAL TRIAL: NCT07038707
Title: Research on the Identification of Early Screening Markers for Herpes Zoster Neuralgia Based on Intestinal Flora Analysis
Brief Title: Early Screening Markers of Herpes Zoster Neuralgia
Status: Not yet recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Xuebi Tian, Clinical Professor, Tongji Hospital
Other Study IDs: TJ-IRB20250519
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Postherpetic Neuralgia ( PHN ); Lymphatic System Disorder
Keywords: Intestinal flora; Inflammation; Lymphatic System Disorder; Postherpetic Neuralgia ( PHN )
MeSH Terms: conditions — Neuralgia, Postherpetic; Lymphatic Diseases; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control group: Healthy individuals matched by age and gender (without a history of HZ or chronic pain diseases).
  Interventions: Other: Extract the serum and feces of the patients for standard screening of early biomarkers; Other: Meningeal lymphatic vessel imaging
- PHN Group: Individuals among patients with herpes zoster (HZ) who eventually develop PHN (according to the diagnostic criteria of PHN, such as persistent pain for ≥3 months)
  Interventions: Other: Extract the serum and feces of the patients for standard screening of early biomarkers; Other: Meningeal lymphatic vessel imaging
- HZ did not convert to the PHN group: Individuals among patients with herpes zoster who did not develop PHN (with complete remission of pain within 3 months).
  Interventions: Other: Extract the serum and feces of the patients for standard screening of early biomarkers; Other: Meningeal lymphatic vessel imaging

INTERVENTIONS:
Other: Extract the serum and feces of the patients for standard screening of early biomarkers — In this study, blood and fecal samples from patients with herpes and herpes neuralgia were collected for genomic sequencing of the gut microbiota and metabolome analysis, etc. Based on the principle of diffusion tensor imaging, by measuring the anisotropic diffusion of white matter around the corpus callosum at the horizontal level of the lateral ventricle body, the lymphatic system clearance function is quantified
Other: Meningeal lymphatic vessel imaging — The functional changes of the cerebral lymphatic system in patients with PHN were detected by meningeal lymphatic vessel imaging

SUMMARY:
Herpes zoster (HZ), especially postherpetic neuralgia, is one of the most typical types of clinical neuralgia. The incidence rate of HZ in China is approximately 7.7%. Among them, 29.8% of HZ patients eventually develop PHN. About 20% of PHN patients suffer from severe neuralgia for more than one year, or even ten years. It is worth noting that patients with neuralgia are prone to comorbidities such as depression, anxiety and sleep disorders, which seriously affect their work efficiency and quality of life. This is a great torment to both the patients and their families, and it also imposes a heavy burden on the medical system.

Professor Xiao Lizu, a collaborator of our team, has discovered in clinical practice that spinal cord electrical stimulation for HZ patients can significantly reduce the risk of developing PHN. Other therapies for reducing the risk of PHN include multiple parvertebral injections of local anesthetics/steroids, which require patients to return for repeated visits. Although these intervention measures have good effects, they may bring additional economic burdens to patients, treatment side effects and prolong their hospital stays. Therefore, they are not suitable for all patients. From this perspective, our development of early screening methods and selective non-pharmacological intervention only for high-risk patients will improve the overall treatment status of HZ, effectively reduce the incidence of PHN, and alleviate the burden on medical insurance and the medical system at the same time.

This project aims to conduct the following research by analyzing the intestinal flora of patients: identifying biomarkers with the ability to predict the risk of PHN in patients, constructing a machine learning classifier for risk prediction, and developing an early screening kit based on this.

Furthermore, traditional studies mostly focus on a single pathological link and lack systematic multi-dimensional analysis. In recent years, the cerebral lymphatic system, as a key pathway for the clearance of metabolic wastes in the brain, has attracted widespread attention. Furthermore, the role of the gut-brain axis in pain regulation has gradually been recognized. Therefore, it is of great scientific significance to integrate and explore the pathological mechanism of PHN from three dimensions: the lymphatic system, neuroinflammation, and intestinal flora.

This project assumes that patients with PHN have a pathological triad of "lymphoid dysfunction - neuroinflammatory activation - intestinal flora imbalance". The specific manifestations are as follows: Impaired lymphoid clearance function (decreased DTI-ALPS index and increased free water), activated systemic inflammatory response (elevated TNF-α and IL-6), and disordered intestinal flora structure (decreased α diversity and increased opportunistic pathogenic bacteria). The three interact with each other and have a synergistic effect, jointly participating in the pathogenesis of PHN.The expected outcome of this project may provide new options for pain management of the large group of neuralgia patients, improve their quality of life, and has great practicality and practical value.

ELIGIBILITY:
Inclusion Criteria:

* The definite diagnoses were PHN (disease course ≤ 1 month), PHN (1 month < disease course < 2 months), and PHN (disease course > 3 months); Age equal to 50 years old; Not accompanied by other chronic pain diseases; Sign the informed consent form.

Exclusion Criteria:

* There are underlying digestive system diseases such as irritable bowel syndrome and inflammatory bowel disease; There are obvious gastrointestinal discomfort symptoms such as diarrhea and abdominal distension; There is immunosuppression or autoimmune disease; Antibiotics, acid suppressants or drugs that interfere with the intestinal flora have been used within the past month; Have a history of mental illness or abuse of tobacco and alcohol (2 packs per day)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals among patients with herpes zoster (HZ) who eventually develop PHN (according to the diagnostic criteria of PHN, such as persistent pain for ≥3 months)
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
HZ biomarkers | 1 week
  DNA was extracted from fecal samples for metagenomic sequencing. Based on the metagenomic sequencing results, we will select the important biomarkers that can distinguish the subgroups of HZ patients

SECONDARY OUTCOMES:
Lymphatic system function | 1 week
  The lymphatic function of patients with PHN was evaluated through a meningeal lymphatic vessel imaging system